CLINICAL TRIAL: NCT00002528
Title: Surgical Therapy With or Without Axillary Node Clearance for Breast Cancer in the Elderly Who Receive Adjuvant Therapy With Tamoxifen.
Brief Title: Surgery With or Without Lymph Node Removal in Treating Older Women With Stage I or Stage IIA Breast Cancer
Acronym: 10-93
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000078383; IBCSG-10-93; EU-93013; NCI-F93-0008
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery w/ axillary clearance, tamox (Experimental): Either a total mastectomy with axillary clearance, or a lesser procedure (quadrantectomy or lumpectomy with radiotherapy to the conserved breast) with axillary lymph node dissection, and tamoxifen (20 mg) given after surgery for the duration of 5 years or until relapse.
  Interventions: Drug: tamoxifen citrate; Procedure: conventional surgery; Radiation: radiation therapy; Procedure: Axillary clearance
- Surgery w/o axillary clearance, tamox (Experimental): Either a total mastectomy without axillary clearance, or a lesser procedure (quadrantectomy or lumpectomy with radiotherapy to the conserved breast) without axillary lymph node dissection, and tamoxifen (20 mg) given after surgery for the duration of 5 years or until relapse.
  Interventions: Drug: tamoxifen citrate; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: tamoxifen citrate — 20 mg daily beginning within 6 weeks of surgery for 5 years or until relapse, whichever occurs first.
Procedure: conventional surgery — Either total mastectomy or, optionally if the tumor was smaller than 5 cm, a breast conserving procedure (lumpectomy or quadrantectomy).
Radiation: radiation therapy — No radiotherapy is to be given after mastectomy. Radiotherapy is optional after breast conserving surgery according to prospectively determined guidelines within each institution. It should be given to the breast only and not to the draining node areas.
Procedure: Axillary clearance — Axillary node dissection.
  Arms: Surgery w/ axillary clearance, tamox

SUMMARY:
RATIONALE: Removing axillary lymph nodes may be effective in stopping the spread of breast cancer cells. It is not yet known if surgery to remove breast cancer is more effective with or without lymph node removal.

PURPOSE: Randomized phase III trial to compare the effectiveness of breast surgery with or without removal of axillary lymph nodes in treating women who have stage I or stage IIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare local and systemic disease-free survival, ipsilateral axillary relapse, occurrence of postmastectomy syndrome, and overall survival of elderly women with clinically operable stage I or IIA breast cancer who subsequently receive adjuvant tamoxifen after treatment with breast surgery with or without axillary node dissection.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to whether they received prior primary surgery (yes vs no) and participating center.

* Arm I: Patients undergo mastectomy, lumpectomy, or quadrantectomy with axillary clearance. Patients then receive oral tamoxifen for 5 years. Patients may also undergo sentinel node biopsy.
* Arm II: Patients undergo surgery as in arm I without axillary clearance. Patients then receive oral tamoxifen for 5 years.

Patients in both arms who undergo breast-conserving surgery may receive optional radiotherapy for 5-6 weeks to the remaining breast tissue, chest, and lung. Upon recurrence in the conserved breast, patients undergo total mastectomy; those in arm II who experience ipsilateral axillary recurrence undergo surgical excision. Adjuvant tamoxifen and follow up are continued.

Quality of life is assessed.

Patients are followed every 3 months for 1 year, every 6 months while receiving tamoxifen, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,020 patients will be accrued for this study within approximately 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage I or IIA breast carcinoma that is considered operable
* No prior axillary clearance or biopsy
* Complete excisional biopsy of primary tumor without axillary clearance or biopsy allowed
* Suspicious manifestations of metastatic disease (e.g., hot spots on bone scan or skeletal pain of unknown cause) must be proven benign
* No bilateral breast cancer (any mass in contralateral breast must be proven benign by biopsy)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 60 and over

Sex:

* Female

Menopausal status

* Postmenopausal

Performance status:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.1 mg/dL
* AST less than 60 U/L

Renal:

* Creatinine less than 1.3 mg/dL

Cardiovascular:

* Normal cardiac function
* No history of congestive heart failure

Other:

* No nonmalignant systemic disease that would preclude protocol therapy or prolonged follow-up
* No psychiatric or addictive disorder that would preclude protocol therapy or informed consent
* No other prior or concurrent malignancy except nonmelanomatous skin cancer or adequately treated carcinoma in situ of the cervix
* Geographically accessible for follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for breast cancer

Chemotherapy:

* No prior chemotherapy for breast cancer

Endocrine therapy:

* No prior endocrine therapy for breast cancer

Radiotherapy:

* No prior radiotherapy for breast cancer

Surgery:

* See Disease Characteristics

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 1993-05; Primary Completion 2002-12 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 17 years from randomization
  Time from randomization to recurrence, metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | 17 years from randomization
  Time from randomization to death.
Toxicity | 17 years from randomization
  Side effects of treatment, especially surgery-related events.
Quality of life | 17 years from randomization
  Quality of life will be assessed by standard International Breast Cancer Study Group instruments

CONTACTS AND LOCATIONS:
Overall Officials: Diana Crivellari, MD, Study Chair — Centro di Riferimento Oncologico - Aviano
Locations (21):
- Australia (5):
  - Royal Prince Alfred Hospital, Sydney, Sydney, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Anti-Cancer Council of Victoria, Melbourne, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Perth, Perth, Western Australia
- National Institute of Oncology, Budapest, Hungary
- Hadassah University Hospital, Jerusalem, Israel
- Italy (5):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Spedali Civili, Brescia
  - Presidio Ospedaliero-Gorizia, Gorizia
  - Ospedale Civile Rimini, Rimini
  - Ospedale San Eugenio, Rome
- Auckland Adventist Hospital, Auckland, New Zealand
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia
- Groote Schuur Hospital, Cape Town, Cape Town, South Africa
- Sahlgrenska University Hospital, Gothenburg (Goteborg), Sweden
- Switzerland (5):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - UniversitaetsSpital, Zurich

REFERENCES:
- [Background] Pestalozzi BC, Zahrieh D, Mallon E, Gusterson BA, Price KN, Gelber RD, Holmberg SB, Lindtner J, Snyder R, Thurlimann B, Murray E, Viale G, Castiglione-Gertsch M, Coates AS, Goldhirsch A; International Breast Cancer Study Group. Distinct clinical and prognostic features of infiltrating lobular carcinoma of the breast: combined results of 15 International Breast Cancer Study Group clinical trials. J Clin Oncol. 2008 Jun 20;26(18):3006-14. doi: 10.1200/JCO.2007.14.9336. Epub 2008 May 5. PMID 18458044
- [Result] International Breast Cancer Study Group; Rudenstam CM, Zahrieh D, Forbes JF, Crivellari D, Holmberg SB, Rey P, Dent D, Campbell I, Bernhard J, Price KN, Castiglione-Gertsch M, Goldhirsch A, Gelber RD, Coates AS. Randomized trial comparing axillary clearance versus no axillary clearance in older patients with breast cancer: first results of International Breast Cancer Study Group Trial 10-93. J Clin Oncol. 2006 Jan 20;24(3):337-44. doi: 10.1200/JCO.2005.01.5784. Epub 2005 Dec 12. PMID 16344321